CLINICAL TRIAL: NCT01153568
Title: Vitamin D and Osteoporosis Prevention in Elderly African American Women: A 4-year Randomized, Double-blind, Placebo-controlled Study to Investigate the Effect of Vitamin D Status in Elderly African American Women
Brief Title: Vitamin D and Osteoporosis Prevention in Elderly African American Women
Acronym: NIHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Winthrop University Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, John F. Aloia, MD, Chief Academic Officer, Winthrop University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 08032; R01AG032440 (NIH)
Record Dates: First submitted 2010-06-28; First posted 2010-06-30 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-06

CONDITIONS: Determine Effect of Vitamin D on Bone Health in Elderly African American Women
Keywords: Vitamin D; osteoporosis; african american women
MeSH Terms: conditions — Osteoporosis | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): placebo
  Interventions: Other: placebo
- Vitamin D 3 (Experimental): Vitamin D3 will be available in doses of 60, 90, 120, and 150 µg
  Interventions: Dietary Supplement: Vitamin D 3

INTERVENTIONS:
Dietary Supplement: Vitamin D 3 — Patients will bew given a single capsule to take once daily
  Arms: Vitamin D 3
Other: placebo — placebo tablets
  Arms: Placebo

SUMMARY:
Vitamin D is a hormone that is produced when sunlight is absorbed by the skin. Vitamin D insufficiency has been recognized as a problem in areas where sun exposure is limited, especially in the wintertime. In addition, the more pigmented the skin is, the less capable it is of utilizing sunlight to make vitamin D. Vitamin D plays an important role in helping the body absorb calcium and in building strong bones. It has also been shown to improve muscle function in the elderly. As we get older, our vitamin D levels in the blood go down and this may increase the risk for falls and fractures. If we can improve vitamin D status as we age, we may be able to improve muscle strength and decrease the risk of falls and fractures.

DETAILED DESCRIPTION:
The long-term goal of this project is to develop strategies for the prevention of osteoporotic fractures in African Americans. Most intervention studies have excluded African Americans because of the erroneous belief that osteoporosis is not a major health problem in this population. In fact, the incidence rate of hip fracture in blacks is 50% of the rate in whites. Since longevity is increasing in the black population, osteoporotic fractures will become an even greater problem for this ethnic minority in the future. Furthermore, morbidity and mortality from osteoporotic fractures is greater in blacks. The elderly require higher intake of vitamin D to prevent bone loss resulting from secondary hyperparathyroidism. Calcium with sufficient vitamin D supplementation may decrease fractures in elderly white populations as a result of reduction in bone loss and falls (improved physical performance). The only fracture intervention study to include African Americans-the Women's Health Initiative-used an inadequate dose of vitamin D (400 IU), a dose unlikely to achieve the vitamin D status proposed by U.S. experts: serum 25 hydroxyvitamin D [25(OH)D] concentration above 75 nmol/L. No calcium/vitamin D intervention studies on fall prevention or physical performance have included African Americans.

As a result of increased skin pigmentation, blacks synthesize less vitamin D from sun exposure. As a result, serum 25(OH)D levels are often in the "insufficient" range. This is accompanied by secondary hyperparathyroidism, but adult blacks have a relative skeletal resistance to PTH, so that they have lower bone turnover. They also have more efficient renal conservation of calcium starting in childhood. Addition of vitamin D3 to a calcium-sufficient African American postmenopausal population does not prevent bone loss. The calcium/vitamin D requirements of black adults may be lower than white adults through midlife. However, the elderly require more vitamin D to produce the higher 25(OH)D levels required to overcome the hyperparathyroidism associated with aging. The skeleton of elderly African Americans appears to be susceptible to the increasing parathyroid hormone levels of old age. Bone loss accelerates and bone turnover markers increase in elderly African Americans just as in whites. The specific aims of this project are to determine if dietary supplementation with calcium/vitamin D will safely reduce bone loss and bone turnover and improve physical performance in elderly African Americans. We will enroll 250 African American women in a four-year vitamin D3 intervention trial where serum 25(OH)D will be maintained at an optimum level above 75 nmol/L. Adequate calcium intake will be ensured. Functional markers of vitamin D including bone density, serum PTH, and bone turnover will be measured. The NIH Conference on Vitamin D and Health in the 21st Century, September 5-6, 2007 concluded that research in this population is a high priority.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory women older than 60 years of age. Self declared as African Americans.
2. 20 nmol/L < serum 25(OH)D level < 65 nmol/L.
3. Willingness to take study drug and participate for four years in the trial.
4. Willingness to refrain from the use of self-administered supplements during the trial.

Exclusion Criteria:

1. Serum 25(OH)D levels ≤ 20 nmol/L or ≥ 65 nmol/L.
2. BMD total hip below - 2.5 standard deviation (using NHANES III adult young white men and women as the point of reference) or history of osteoporotic fracture.
3. Moderate to severe fracture in one or more vertebrae by Instant Vertebral Assessment on DXA.
4. Treatment with HRT, SERMS, calcitonin, PTH, androgens, bisphosphonates, phosphate or anabolic steroids during 6 months prior to entry.
5. Use of systemic corticosteroids (oral or IV) within the last year at an average dose of greater than 5 mg per day of oral prednisone or equivalent for a period of three months or more prior to screening.
6. Hypercalcemia (serum calcium > 10.6 mg (dl) or history of primary hyperparathyroidism.
7. History of chronic liver disease, chronic renal insufficiency, Parkinson's, metabolic bone disease, hematologic tumors, rheumatologic disease requiring steroids, malabsorption or new diagnosis or active treat-ment of cancer 12 months prior to inclusion.
8. Use of medications that influence bone metabolism (e.g. anticonvulsants).
9. Significant deviation from normal in either: history, physical examination or laboratory tests as evaluated by the Principle Investigator. Participants with a history of hypercalciuria, nephrolithiasis and active sarcoidosis will also be excluded.
10. Participation in another investigational trial 30 days prior to screening.
11. Spinal disease that affects interpretation of bone densitometry like scoliosis with a Cobb angle greater than 15o, history of surgery at lumbosacral spine.
12. Bilateral hip replacement.
13. Currently smoking more than 10 cigarettes daily.
14. Body width on DXA > 25 cm.
15. Patients who are deemed unsafe to perform muscular function testing as evaluated by the investigator.

    ---------- Study participants should live close to the study site, as this study requires multiple visits over a four year period.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2010-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
1. To determine if vitamin D supplementation sufficient to raise serum 25(OH)D levels above 75 nmol/L (30 ng/mL) for four years will reduce bone density loss, markers of bone turnover, and serum PTH in elderly black women | 4 years
  2. To determine whether such supplementation will inhibit the decline in physical performance with aging.

SECONDARY OUTCOMES:
To evaluate the harms of vitamin D intakes that raise 25(OH)D levels above 75 nmol/L for four years in a calcium sufficient population | 4 years
  This research will fill an important gap in knowledge about the potential benefit of vitamin D supplementation in elderly black women. While many experts agree that vitamin D intake should be increased in the elderly, few pertinent studies have included black participants, who represent a vulnerable population due to their low serum 25(OH)D. If vitamin D supplementation proves to be beneficial in this minority group, that would suggest the appropriateness of intake recommendations similar to those proposed for white populations.

CONTACTS AND LOCATIONS:
Overall Officials: John F. Aloia, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States

REFERENCES:
- [Background] Bischoff-Ferrari HA, Giovannucci E, Willett WC, Dietrich T, Dawson-Hughes B. Estimation of optimal serum concentrations of 25-hydroxyvitamin D for multiple health outcomes. Am J Clin Nutr. 2006 Jul;84(1):18-28. doi: 10.1093/ajcn/84.1.18. PMID 16825677
- [Background] Aloia JF, Vaswani A, Yeh JK, Flaster E. Risk for osteoporosis in black women. Calcif Tissue Int. 1996 Dec;59(6):415-23. doi: 10.1007/BF00369203. PMID 8939764
- [Background] Cauley JA, Lui LY, Stone KL, Hillier TA, Zmuda JM, Hochberg M, Beck TJ, Ensrud KE. Longitudinal study of changes in hip bone mineral density in Caucasian and African-American women. J Am Geriatr Soc. 2005 Feb;53(2):183-9. doi: 10.1111/j.1532-5415.2005.53101.x. PMID 15673339
- [Background] Tang BM, Eslick GD, Nowson C, Smith C, Bensoussan A. Use of calcium or calcium in combination with vitamin D supplementation to prevent fractures and bone loss in people aged 50 years and older: a meta-analysis. Lancet. 2007 Aug 25;370(9588):657-66. doi: 10.1016/S0140-6736(07)61342-7. PMID 17720017
- [Background] Vieth R, Ladak Y, Walfish PG. Age-related changes in the 25-hydroxyvitamin D versus parathyroid hormone relationship suggest a different reason why older adults require more vitamin D. J Clin Endocrinol Metab. 2003 Jan;88(1):185-91. doi: 10.1210/jc.2002-021064. PMID 12519850
- [Background] Bischoff-Ferrari HA, Willett WC, Wong JB, Giovannucci E, Dietrich T, Dawson-Hughes B. Fracture prevention with vitamin D supplementation: a meta-analysis of randomized controlled trials. JAMA. 2005 May 11;293(18):2257-64. doi: 10.1001/jama.293.18.2257. PMID 15886381
- [Background] Latham NK, Anderson CS, Lee A, Bennett DA, Moseley A, Cameron ID; Fitness Collaborative Group. A randomized, controlled trial of quadriceps resistance exercise and vitamin D in frail older people: the Frailty Interventions Trial in Elderly Subjects (FITNESS). J Am Geriatr Soc. 2003 Mar;51(3):291-9. doi: 10.1046/j.1532-5415.2003.51101.x. PMID 12588571
- [Background] MacLaughlin J, Holick MF. Aging decreases the capacity of human skin to produce vitamin D3. J Clin Invest. 1985 Oct;76(4):1536-8. doi: 10.1172/JCI112134. PMID 2997282
- [Background] Dawson-Hughes B, Heaney RP, Holick MF, Lips P, Meunier PJ, Vieth R. Estimates of optimal vitamin D status. Osteoporos Int. 2005 Jul;16(7):713-6. doi: 10.1007/s00198-005-1867-7. Epub 2005 Mar 18. PMID 15776217
- [Background] Vieth R, Bischoff-Ferrari H, Boucher BJ, Dawson-Hughes B, Garland CF, Heaney RP, Holick MF, Hollis BW, Lamberg-Allardt C, McGrath JJ, Norman AW, Scragg R, Whiting SJ, Willett WC, Zittermann A. The urgent need to recommend an intake of vitamin D that is effective. Am J Clin Nutr. 2007 Mar;85(3):649-50. doi: 10.1093/ajcn/85.3.649. No abstract available. PMID 17344484
- [Background] Visser M, Deeg DJ, Puts MT, Seidell JC, Lips P. Low serum concentrations of 25-hydroxyvitamin D in older persons and the risk of nursing home admission. Am J Clin Nutr. 2006 Sep;84(3):616-22; quiz 671-2. doi: 10.1093/ajcn/84.3.616. PMID 16960177
- [Background] Dhesi JK, Bearne LM, Moniz C, Hurley MV, Jackson SH, Swift CG, Allain TJ. Neuromuscular and psychomotor function in elderly subjects who fall and the relationship with vitamin D status. J Bone Miner Res. 2002 May;17(5):891-7. doi: 10.1359/jbmr.2002.17.5.891. PMID 12009020
- [Background] Bischoff HA, Stahelin HB, Dick W, Akos R, Knecht M, Salis C, Nebiker M, Theiler R, Pfeifer M, Begerow B, Lew RA, Conzelmann M. Effects of vitamin D and calcium supplementation on falls: a randomized controlled trial. J Bone Miner Res. 2003 Feb;18(2):343-51. doi: 10.1359/jbmr.2003.18.2.343. PMID 12568412
- [Background] Wicherts IS, van Schoor NM, Boeke AJ, Visser M, Deeg DJ, Smit J, Knol DL, Lips P. Vitamin D status predicts physical performance and its decline in older persons. J Clin Endocrinol Metab. 2007 Jun;92(6):2058-65. doi: 10.1210/jc.2006-1525. Epub 2007 Mar 6. PMID 17341569
- [Background] Bischoff-Ferrari HA, Dawson-Hughes B, Willett WC, Staehelin HB, Bazemore MG, Zee RY, Wong JB. Effect of Vitamin D on falls: a meta-analysis. JAMA. 2004 Apr 28;291(16):1999-2006. doi: 10.1001/jama.291.16.1999. PMID 15113819
- [Result] Barrett-Connor E, Siris ES, Wehren LE, Miller PD, Abbott TA, Berger ML, Santora AC, Sherwood LM. Osteoporosis and fracture risk in women of different ethnic groups. J Bone Miner Res. 2005 Feb;20(2):185-94. doi: 10.1359/JBMR.041007. Epub 2004 Oct 18. PMID 15647811
- [Derived] Aloia JF, Islam S, Mikhail M. Vitamin D and Acute Respiratory Infections-The PODA Trial. Open Forum Infect Dis. 2019 Sep 4;6(9):ofz228. doi: 10.1093/ofid/ofz228. eCollection 2019 Sep. PMID 31660391
- [Derived] Aloia JF, Mikhail M, Fazzari M, Islam S, Ragolia L, Guralnik J. Physical Performance and Vitamin D in Elderly Black Women-The PODA Randomized Clinical Trial. J Clin Endocrinol Metab. 2019 May 1;104(5):1441-1448. doi: 10.1210/jc.2018-01418. PMID 30496578
- [Derived] Aloia J, Fazzari M, Islam S, Mikhail M, Shieh A, Katumuluwa S, Dhaliwal R, Stolberg A, Usera G, Ragolia L. Vitamin D Supplementation in Elderly Black Women Does Not Prevent Bone Loss: A Randomized Controlled Trial. J Bone Miner Res. 2018 Nov;33(11):1916-1922. doi: 10.1002/jbmr.3521. Epub 2018 Jul 19. PMID 29905969
- See also: National Osteoporosis Foundation — http://www.nof.org
- See also: National Institute of Arthritis and Musculoskeletal and Skin Diseases — http://www.niams.nih.gov